CLINICAL TRIAL: NCT02239146
Title: A Multi-Centre, Randomised, Double-Blind, Placebo Controlled, Dose Escalation Trial on Safety and Pharmacokinetics of Recombinant Factor XIII (rFXIII) in Patients Following First Time Myocardial Revascularization Requiring Cardiopulmonary Bypass
Brief Title: Safety of rFXIII in Patients Following First Time Myocardial Revascularization Requiring Cardiopulmonary Bypass
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Novo Nordisk A/S (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: F13CARD-1660; 2005-000729-40 (EudraCT Number)
Record Dates: First submitted 2014-09-10; First posted 2014-09-12 (Estimated); Last update posted 2017-01-11 (Estimated); Status verified 2017-01

CONDITIONS: Acquired Bleeding Disorder; Cardiac Surgery Requiring Cardiopulmonary Bypass

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- rFXIII (Experimental)
  Interventions: Drug: catridecacog
- Placebo (Placebo Comparator)
  Interventions: Drug: placebo

INTERVENTIONS:
Drug: catridecacog — Single doses of rFXIII administered intravenously (i.v.) to eight subjects in each of the four dose groups (11.9, 25, 35 and 50 IU/kg).
  Arms: rFXIII
Drug: placebo — Single doses of placebo administered intravenously (i.v.) to two subjects in each of the four dose groups (11.9, 25, 35 and 50 IU/kg).
  Arms: Placebo

SUMMARY:
This trial is conducted in Europe and the United States of America (USA). The aim of this trial is to evaluate the safety of escalating single doses of rFXIII (recombinant factor XIII, catridecacog) administered following first time myocardial revascularization requiring cardiopulmonary bypass (CPB).

ELIGIBILITY:
Inclusion Criteria:

* Subject is undergoing his/her first myocardial revascularization

Exclusion Criteria:

* Previous participation (randomisation and dosing) in this trial
* Subject has a history of cerebrovascular event (including thrombotic or haemorrhagic stroke or transient ischaemic attack (TIA)) and/or extra-myocardial thromboembolic events, e.g., deep vein thrombosis (DVT) or pulmonary embolus (PE)
* Subject required a pre-operative (within 30 days) transfusion of any blood and/or blood product
* Subject has a current atrial fibrillation or history of atrial fibrillation

Ages: 35 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 43 (Actual)
Dates: Start 2005-10; Primary Completion 2008-01 (Actual); Study Completion 2008-01 (Actual)

PRIMARY OUTCOMES:
Incidence and severity of adverse events | From dosing up to 5-7 weeks ± 3 days after trial product administration

SECONDARY OUTCOMES:
Incidence and magnitude of laboratory abnormalities following administration of rFXIII | From dosing up to 5-7 weeks ± 3 days after trial product administration
Incidence of antibodies to FXIII-A subunit | From dosing up to 5-7 weeks ± 3 days after trial product administration
Incidence of anti-yeast antibodies | From dosing up to 5-7 weeks ± 3 days after trial product administration

CONTACTS AND LOCATIONS:
Overall Officials: Global Clinical Registry (GCR, 1452), Study Director — Novo Nordisk A/S
Locations (22):
- United States (13):
  - Novo Nordisk Investigational Site, Tucson, Arizona
  - Novo Nordisk Investigational Site, San Francisco, California
  - Novo Nordisk Investigational Site, Denver, Colorado
  - Novo Nordisk Investigational Site, Indianapolis, Indiana
  - Novo Nordisk Investigational Site, Camden, New Jersey
  - Novo Nordisk Investigational Site, New York, New York
  - Novo Nordisk Investigational Site, The Bronx, New York
  - Novo Nordisk Investigational Site, Cleveland, Ohio
  - Novo Nordisk Investigational Site, Portland, Oregon
  - Novo Nordisk Investigational Site, Allentown, Pennsylvania
  - Novo Nordisk Investigational Site, Philadelphia, Pennsylvania
  - Novo Nordisk Investigational Site, Houston, Texas
  - Novo Nordisk Investigational Site, Richmond, Virginia
- Novo Nordisk Investigational Site, Toronto, Canada
- Novo Nordisk Investigational Site, København Ø, Denmark
- Germany (3):
  - Novo Nordisk Investigational Site, Hamburg
  - Novo Nordisk Investigational Site, Lahr
  - Novo Nordisk Investigational Site, Mainz
- United Kingdom (4):
  - Novo Nordisk Investigational Site, Cambridge
  - Novo Nordisk Investigational Site, London
  - Novo Nordisk Investigational Site, Middlesbrough
  - Novo Nordisk Investigational Site, Southampton

REFERENCES:
- [Result] Levy JH, Gill R, Nussmeier NA, Olsen PS, Andersen HF, Booth FV, Jespersen CM. Repletion of factor XIII following cardiopulmonary bypass using a recombinant A-subunit homodimer. A preliminary report. Thromb Haemost. 2009 Oct;102(4):765-71. doi: 10.1160/TH08-12-0826. PMID 19806264
- See also: Clinical Trials at Novo Nordisk — http://novonordisk-trials.com